CLINICAL TRIAL: NCT01251107
Title: Prospective Randomized Comparison of ABVD Versus BEACOPP Chemotherapy With or Without Radiotherapy for Advanced Stage or Unfavorable Hodgkin's Lymphoma (HL)
Brief Title: Study Comparing ABVD vs BEACOPP in Advanced Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Michelangelo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41/99
Record Dates: First submitted 2010-11-26; First posted 2010-12-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2011-02

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; ABVD; BEACOPP; Salvage high dose chemotherapy
MeSH Terms: conditions — Hodgkin Disease | interventions — Bleomycin; Etoposide; Doxorubicin; Cyclophosphamide; Vincristine; Procarbazine; Prednisone; deltacortene; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm B (Experimental): BEACOPP (Bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, prednisone) for 4 escalated cycles followed by 4 standard cycles
  Interventions: Drug: Bleomycin; Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Procarbazine; Drug: Prednisone
- Arm A (Active Comparator): ABVD (doxorubicin, bleomycin, vinblastine, dacarbazine) for 6 to 8 cycles
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Bleomycin — 10 mg/m2 IV day 8 during cycles 1 to 8
  Other Names: Bleomicina Teva
  Arms: Arm B
Drug: Etoposide — 200 mg/m2 iv on days 1 to 3 during cycles 1 to 4; 100 mg/m2 iv on days 1 to 3 during cycles 5 to 8
  Other Names: VP-16, Etoposide Teva
  Arms: Arm B
Drug: Doxorubicin — 35 mg/2 iv on day 1 during cycles 1 to 4; 25 mg/m2 iv on day 1 during cycles 5 to 8
  Other Names: Adriblastina Pfizer
  Arms: Arm B
Drug: Cyclophosphamide — 1250 mg/m2 iv on day 1 during cycles 1 to 4; 650 mg/m2 iv on day 1 during cycles 5 to 8
  Other Names: Endoxan Baxter
  Arms: Arm B
Drug: Vincristine — 1.4 mg/m2 iv (max 2 mg) on day 8 during cycles 1 to 8
  Other Names: Vincristina Teva Italia
  Arms: Arm B
Drug: Procarbazine — 100 mg/m2 po from day 1 to 7 during cycles 1 to 8
  Other Names: Natulan
  Arms: Arm B
Drug: Prednisone — 40 mg/m2 po from day 1 to 14 during cycles 1 to 8
  Other Names: Deltacortene
  Arms: Arm B
Drug: Doxorubicin — 25 mg/m2 iv on days 1 and 15 in each cycle
  Other Names: Adriblastina Pfizer
  Arms: Arm A
Drug: Bleomycin — 10 mg/m2 iv on days 1 and 15 in each cycle
  Other Names: Bleomicina Teva
  Arms: Arm A
Drug: Vinblastine — 6 mg/m2 iv on days 1 and 15 in each cycle
  Other Names: Velbe
  Arms: Arm A
Drug: Dacarbazine — 375 mg/m2 iv on days 1 and 15 in each cycle
  Other Names: Dacarbazina Medac
  Arms: Arm A

SUMMARY:
The choice of a preferred first-line treatment requires balancing the desire for optimal disease control with the occurrence of early and late treatment-related effects. To fully assess this balance, the treatment decision process should ideally take into account the outcome following a consistent second-line therapy, in particular when tolerated, widely applicable and highly effective salvage regimens exist, like in Hodgkin lymphoma failing initial chemotherapy.

DETAILED DESCRIPTION:
During the last two decades ABVD (doxorubicin, bleomycin, vinblastine, dacarbazine) has been considered as the standard of care for advanced HL, however 20-30% of the patients fail to achieve a durable complete remission and need a salvage treatment. After a state-of-the art-salvage program including high-dose chemotherapy and autologous hematopoietic stem cell support (ASCT) at least half of these patients achieve a durable disease control. Recently the German Hodgkin Study Group (GHSG) has developed a new regimen, BEACOPP (bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine and prednisone), administered with or without dose escalation. In an interim analysis after 23 months follow-up, BEACOPP demonstrated a higher activity compared to COPP/ABVD with a superior freedom from treatment failure (84% versus 75%, P=.034). Despite the improved efficacy a substantial proportion of patients receiving escalated BEACOPP experienced severe acute hematologic toxicity (grade 3-4 leucopoenia, thrombocytopenia and anemia occurred in 78% , 36% and 27% of the cycles administered, respectively) and 1.8% fatal acute toxicities were reported. Moreover of greater concern is the incidence of almost fatal secondary acute leukemia and myelodysplastic syndrome (3 cases in 323 patients). The choice of first-line treatment requires balancing the desire for optimal disease control with the occurrence of early and late treatment-related toxicities. Long-term outcome following an optimal salvage treatment, consisting in high-dose chemotherapy with ASCT should also be taken into consideration. In the present study we plan to compare the efficacy and toxicity of two therapeutic strategies consisting in two different first-line treatments followed by a pre-planned salvage program, when indicated

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed Hodgkin's lymphoma (pathological review diagnosis available)
* No prior treatment
* Stage II B, III A and B, IV A and B
* Normal hematopoietic function as measured by leucocytes equal to or greater than 3500/mm3, neutrophils equal to or greater than 1500/mm3, platelets equal to or greater than 100000/mm3
* Normal renal function (serum creatinine < 1,5x ULN) and normal liver function (SGOT/SGPT equal to or lower than 2.5x ULN; bilirubin equal to or lower than 1.5x ULN)
* No significant history or current evidence of cardiovascular disease, or major respiratory disease
* No severe neurologic or psychiatric disease
* No other malignancy except basal cell carcinoma of the skin and/or in situ cervical carcinoma of the uterus
* Serological negativity for hepatitis B or C or HIV infection
* ECOG performance status equal to or lower than 2
* Life expectancy of at least three months
* Effective contraception in all patients and a negative pregnancy test for women of childbearing potential
* Written informed consent and consent to a regular follow-up in the outpatient clinic

Exclusion criteria:

* Sever central nervous system or psychiatric disease
* History or current evidence of clinically significant cardiac disease (congestive heart failure, uncontrolled hypertension, unstable coronary artery disease or myocardial infarction or severe arrhythmias. Left ventricular ejection fraction < 50% at rest by echocardiography or < 55% by isotopic measurement
* Serological positivity for HBV, HCV or HIV
* History or current evidence of malignancy other than basal cell carcinoma of the skin, carcinoma in situ of the cervix
* Lactating or pregnant women

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 331 (Actual)
Dates: Start 2000-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Freedom from first progression at 5 years | After a median of 5 years from start of the study

SECONDARY OUTCOMES:
Freedom from second progression at 5 years | After a median of 5 years from start of protocol
Overall survival at 5 years | After a median of 5 years from start of the protocol
Number of participants with acute adverse events at initial therapy and at salvage therapy as a measure of safety and tolerability | After 3 months from last intervention
Number of participants long term sequelae | After a median of 10 years
  Number of participants who developed leukemia Number of participants who developed solid tumors Number of participants who developed cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro M Gianni, MD, Study Chair — Fondazione IRCCS Istituto Nazionale Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale di Tumori di Milano, Milan, Italy

REFERENCES:
- [Derived] Viviani S, Zinzani PL, Rambaldi A, Brusamolino E, Levis A, Bonfante V, Vitolo U, Pulsoni A, Liberati AM, Specchia G, Valagussa P, Rossi A, Zaja F, Pogliani EM, Pregno P, Gotti M, Gallamini A, Rota Scalabrini D, Bonadonna G, Gianni AM; Michelangelo Foundation; Gruppo Italiano di Terapie Innovative nei Linfomi; Intergruppo Italiano Linfomi. ABVD versus BEACOPP for Hodgkin's lymphoma when high-dose salvage is planned. N Engl J Med. 2011 Jul 21;365(3):203-12. doi: 10.1056/NEJMoa1100340. PMID 21774708